CLINICAL TRIAL: NCT01563627
Title: Serum Profile of Inflammatory Factors, Immune and Angiogenic in Temporal Lobe Epilepsy: New Targets for Diagnosis and Prediction of Drug Resistance
Brief Title: Serum Profile of Inflammatory Factors, Immune and Angiogenic in Temporal Lobe Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 8668
Record Dates: First submitted 2012-03-09; First posted 2012-03-27 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Blood Specimen Collection; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antiepileptic Drug resistant (Experimental): Adult patients suffering from epilepsy drug-resistant and potentially surgical candidates
  Interventions: Other: blood sampling for drug resistance biomarkers; Device: Magnetic Resonance Imaging
- Antiepileptic drug Controlled group (Experimental): epilepsy well controlled by antiepileptic drugs
  Interventions: Other: blood sampling for drug resistance biomarkers; Device: Magnetic Resonance Imaging

INTERVENTIONS:
Other: blood sampling for drug resistance biomarkers — comparison of Inflammatory Factors, Immune and Angiogenic in Temporal Lobe Epilepsy
Device: Magnetic Resonance Imaging

SUMMARY:
Epilepsy affects 0.7% of the general population and 15-20% of patients develop drug resistance. The temporal lobe epilepsy (TLE) is the most common symptomatic focal epilepsies with a particularly high rate of drug (about 20 to 30%). In this type of epilepsy, where feasible, surgical removal of the home is the best therapeutic outcome.

Mechanisms of epileptogenesis and drug resistance are still mysterious. Of recent clinical and experimental studies have shown that dysfunction of the blood-brain barrier (BBB) contributes to epileptogenesis and drug resistance. It is now recognized that cytokines exacerbate the excitability and permeability of the BBB, which was recently confirmed by studies showing that treatment of inflammation reduces epileptogenesis. Moreover, we have described an association between pathological angiogenesis and BBB permeability in the tissue of patients with excision of drug-resistant TLE. With experimental models, it was revealed an activation of the VEGF-VEGFR2 by seizures leading to rapid degradation of the BBB.

The investigators hypothesis is that the identification of factors involved in BBB permeability may designate potential targets for drug-resistant partial epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with temporal lobe epilepsy (TLE)
* Patient with epilepsy for at least two years. Arm 1: Patient with drug-resistant TLE proved potentially a candidate for surgery.

Arm 2: Patient with TLE seizure-free for 12 months or more

Exclusion Criteria:

* Patient with a scalable general pathology may lead to increased inflammatory markers: neoplasia, chronic inflammatory diseases etc. ...
* Patient with neurological history other than epilepsy with evolutionary potential or likely to interfere with the inflammatory markers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Comparison of Biomarkers | 12 months after inclusion (day 0)
  Identify blood sampling biomarkers of drug resistance in temporal lobe epilepsy, an analysis by large-scale expression profiling of serum factors involved in inflammation, immunity and angiogenesis

SECONDARY OUTCOMES:
permeability of the blood-brain barrier | Day 0
  Compare changes in lesion morphologic imaging and blood flow measurements by Magnetic Resonance Imaging between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- UH Montpellier, Montpellier, France